CLINICAL TRIAL: NCT03365492
Title: BioFreedom PK Study in Patients With CAD Who Receive the BioFreedom™ Biolimus A9™ Stent
Brief Title: BioFreedom Pharmacokinetic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17EU03
Record Dates: First submitted 2017-11-23; First posted 2017-12-07 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Commercially available BioFreedomTM (stainless steel BA9TM drug-coated stent)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with CAD who receive the BioFreedom™ Biolimus A9™ stent.
  Interventions: Device: BioFreedom™ BA9™ drug-coated stent

INTERVENTIONS:
Device: BioFreedom™ BA9™ drug-coated stent — Drug-coated stent for coronary arteries

SUMMARY:
The purpose of this pharmacokinetic (PK) study is to characterize the maximum concentration (Cmax) and time-to-maximum concentration (Tmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus in a cohort of coronary artery disease (CAD) patients following implantation of BioFreedomTM SS stent.

DETAILED DESCRIPTION:
The purpose of this pharmacokinetic (PK) study is to characterize the maximum concentration (Cmax) and time-to-maximum concentration (Tmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus in a cohort of coronary artery disease (CAD) patients following implantation of BioFreedomTM SS stent.

The study will include up to 20 CAD patients following implantation of the commercially available BioFreedomTM SS stent in a single Spanish center. Venous blood samples will be taken up to 72 hours after implantation. Whole blood concentrations of Biolimus A9TM and its active metabolites sirolimus and everolimus will be determined using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) assay. Mean, median and range of PK variables (Cmax, Tmax, and AUC) together with a Summary Statistics table will be generated as part of the PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Symptomatic coronary artery disease including patients with chronic stable angina, unstable angina, silent ischemia, and acute coronary syndromes including non-ST elevation myocardial infarction;
3. Presence of one or more coronary artery stenoses >50% in a native coronary artery from 2.25 to 4.0 mm in diameter that can be covered with one or more stents;
4. Patient receives one or more BioFreedom stents resulting in a total stent length ranging from 30mm to 45mm;

Exclusion Criteria:

1. Individual is pregnant, nursing or planning to be pregnant;
2. Patient presents with STEMI;
3. Known intolerance to aspirin, clopidogrel, heparin, zinc, stainless steel, Biolimus A9TM or contrast material;
4. Inability to provide informed consent;
5. Currently participating in another trial;
6. Treatment with any DES within the previous 6 months;
7. Patient requires a stent <2.25mm;
8. Patient requires a stent >4.0mm;
9. Patient receives a non-study DES stent during the index procedure;
10. Use of a drug coated balloon planned at the index procedure;
11. Systemic use of a -limus drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
To characterize the maximum concentration (Cmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus | Measured upto 72 hours after stent implantation
  To characterize the maximum concentration (Cmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus
To characterize the time-to-maximum concentration (Tmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus | Measured upto 72 hours after stent implantation
  To characterize the time-to-maximum concentration (Tmax) of Biolimus A9TM and its active metabolites sirolimus and everolimus

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain